CLINICAL TRIAL: NCT03645694
Title: Social Support Aid For People With Dementia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Advanced Medical Electronics (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1502S63961; R44AG041667 (NIH)
Record Dates: First submitted 2018-08-17; First posted 2018-08-24 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Dementia; Memory Loss
Keywords: Caregiving; Technology; Social support
MeSH Terms: conditions — Dementia; Memory Disorders

STUDY DESIGN:
Intervention Model Description: Individual with memory concerns and their family caregivers were randomly assigned to receive the facial recognition technology or usual care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SSA (Experimental): Individuals with memory concerns in the experimental arm received the prototype facial recognition technology, which included a smartphone and smartwatch. The smartphone was equipped with facial recognition software application; the smartwatch communicated information with the smartphone. Persons with memory concerns and their family care partners were given a demonstration on how to utilize the technology.
  Interventions: Device: Social Support Aid
- Control (No Intervention): Control participants did not receive the technology; at the conclusion of follow-up, all controls were offered the technology to use.

INTERVENTIONS:
Device: Social Support Aid — Please see earlier; the social support aid technology consists of a smartphone with a facial recognition software application and a smartwatch. Up to 1,000 individuals can be enrolled in the facial recognition application. Enrollment includes typing individuals names and relationships of the person with memory concern into the application and taking pictures of PWMC's faces at multiple angles. Once enrolled and in view of the smartphone's camera, the SSA's application recognizes the individual's face and alerts the smartwatch. The watch then vibrates and displays the individuals' name and relationship to the PWMC.
  Arms: SSA

SUMMARY:
The goal of this study is to determine the acceptability, utility, and preliminary effectiveness of a facial recognition technology for persons with memory concerns and their family care partners.

DETAILED DESCRIPTION:
This project develops a novel social support aid (SSA) to allow persons with memory concerns (PWMCs) to more fully engage in their social network and enhance their quality of life. The SSA will assist people in an early stage of dementia, e.g., Alzheimer's disease or related dementia, who desire social interaction, but struggle to remember names and relationships. It provides memory cuing by displaying the names and relationships of the people with whom PWMCs are engaged. The investigators anticipate that the SSA will offer robust support for care partners and PWMCs in various communities. The SSA is not intended to replace caregiver aids, but rather augment them to further improve quality of life. Millions of Americans have dementia, the loss of mental functions, e.g., thinking, memory, and reasoning, which interferes with their daily functioning. While some cases of dementia are caused by medical conditions that can be treated, most cannot be reversed. Hence, the focus switches from treatment to palliative care, i.e., developing a plan to make life easier and more comfortable for individuals with dementia and their caregivers. Assistive technologies to enhance living with dementia, let alone studies that evaluate their efficacy, are underdeveloped. The proposed project aims to begin filling this scientific and clinical gap by developing a social support aid and formally evaluating its utility via a sufficiently powered randomized controlled trial.

This phase II Small Business Innovation Research project will continue work started in phase I and complete a product. The aim of this human subjects research protocol is to evaluate whether the SSA exerts positive benefits for PWMCs' social connections, communication, and quality of life via an embedded experimental mixed methods design that combines the collection and analysis of qualitative data within a traditional randomized controlled trial (RCT) design. The investigators hypothesize that the proposed SSA will exert positive benefits on the social connections, communication, and quality of life of people in early stage dementia.

ELIGIBILITY:
Inclusion Criteria:

PWMCs must be:

* A physician diagnosis of early-stage Alzheimer's disease, mild cognitive impairment, or a self-identified concern of memory loss.
* Able to complete surveys in English or Spanish
* SLUMS score of 20 or above

Care partners of PWMCs must be:

* 21 years of age and over;
* self-identify as someone who provides assistance to the PWMC because of their memory loss (these individuals are called ''care partners,'' as these individuals may or may not provide the intensive hands-on care typical of ''caregivers'');
* indicate a willingness to use the SSA

Exclusion Criteria:

* Indicates an unwillingness to use the SSA.

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
Change in Dementia Quality of Life | Baseline, 3-months, and 6-months
  The 21-item modified Dementia Quality of Life instrument is a self-report survey that assesses various domains of quality of life in the person wtih dementia.
Change in Cantril quality of life ladder | Baseline, 3-months, and 6-months
  The Cantril quality of life ladder is a single item survey that asks respondents to rate their overall quality of life on a scale of 0 (bottom of the latter) to 10 (top of the ladder).

SECONDARY OUTCOMES:
Pleasant events and activities of person with memory concerns | 3-months and 6-months
  The Pleasant Events and Activities-AD Schedule Short Form is a 17-item self-report survey that measures the degree of enjoyment persons with dementia have engaging in a range of activities.
Change in the frequency and quality of social interactions of persons with memory concerns | Baseline, 3-months, and 6-months
  Series of weekly, self-report calendar measures on types and quality of social interactions, developed for this study.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] McCarron HR, Zmora R, Gaugler JE. A Web-Based Mobile App With a Smartwatch to Support Social Engagement in Persons With Memory Loss: Pilot Randomized Controlled Trial. JMIR Aging. 2019 Jun 18;2(1):e13378. doi: 10.2196/13378. PMID 31518270

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-08): https://cdn.clinicaltrials.gov/large-docs/94/NCT03645694/Prot_SAP_000.pdf